CLINICAL TRIAL: NCT00121810
Title: An Open Label, Randomized, Multicenter Study to Evaluate the Efficacy and Safety of Early Calcineurin Inhibitor Withdrawal in Recipients of Primary Renal Allografts Maintained Long-term on Mycophenolate Mofetil (MMF) (CellCept®) and Sirolimus (Rapamune®)
Brief Title: Kidney Spare the Nephron (STN) Study - A Study of CellCept (Mycophenolate Mofetil) and Rapamune (Sirolimus) in Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Disclosures Group, Hoffmann-La Roche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML17140
Record Dates: First submitted 2005-07-15; First posted 2005-07-21 (Estimated); Results first posted 2011-02-24 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Mycophenolic Acid; Adrenal Cortex Hormones; Calcineurin Inhibitors; Sirolimus

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: mycophenolate mofetil [CellCept]; Drug: Corticosteroids; Drug: Sirolimus
- 2 (Active Comparator)
  Interventions: Drug: mycophenolate mofetil [CellCept]; Drug: Corticosteroids; Drug: Calcineurin inhibitors

INTERVENTIONS:
Drug: mycophenolate mofetil [CellCept] — 1.0-1.5 g oral dose twice daily
Drug: Corticosteroids — As prescribed
Drug: Calcineurin inhibitors — As prescribed
  Arms: 2
Drug: Sirolimus — As prescribed
  Arms: 1

SUMMARY:
This 2-arm study recruited kidney transplant patients who were receiving standard care of calcineurin inhibitors (CNIs, tacrolimus or cyclosporine), CellCept (1.0-1.5 g twice daily) and corticosteroids. They were either randomized to continue this regimen, or CNI therapy was discontinued and replaced by sirolimus therapy (in combination with CellCept and corticosteroids). The effect of these 2 regimens on efficacy, safety and kidney function was evaluated. The anticipated time on study treatment was 1-2 years, and the target sample size was 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-75 years of age
* Kidney transplant 30-180 days post-transplantation
* Receipt of cyclosporine or tacrolimus, CellCept, and corticosteroids for greater than 14 days prior to study entry
* No known contraindications to sirolimus

Exclusion Criteria:

* Multiple organ transplant recipients or secondary kidney transplant recipients
* Corticosteroid-resistant rejection episode within 90 days prior to study entry or corticosteroid-sensitive rejection episode within 30 days prior to study entry
* More than 1 biopsy-proven episode of acute rejection prior to study entry
* Treated with sirolimus before the study
* Organ transplant or expected organ transplant, other than kidney
* History of malignancy in the last 5 years (except successfully treated localized non-melanotic skin cancer)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2003-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (33):
- United States (33):
  - Bakersfield, California
  - Los Angeles, California
  - Palo Alto, California
  - Riverside, California
  - San Diego, California
  - San Francisco, California
  - Denver, Colorado
  - Hartford, Connecticut
  - Washington D.C., District of Columbia
  - Atlanta, Georgia
  - Maywood, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Camden, New Jersey
  - Livingston, New Jersey
  - New York, New York
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Sioux Falls, South Dakota
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Galveston, Texas
  - San Antonio, Texas
  - Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Mycophenolate Mofetil + Sirolimus: Mycophenolate mofetil orally twice daily at a dose of 1.0 g to 1.5 g + sirolimus orally at a dose of 2 g to 10 g followed by a maintenance dose of 2 mg once daily
- Mycophenolate Mofetil + Cyclosporine or Tacrolimus: Mycophenolate mofetil orally twice daily at a dose of 1.0 g to 1.5 g + cyclosporine or tacrolimus according to the study center protocol
Period: Overall Study
Arm/Group | Mycophenolate Mofetil + Sirolimus | Mycophenolate Mofetil + Cyclosporine or Tacrolimus
Started | 151 | 154
Safety Population | 148 | 153
Intent-to-Treat (ITT) Population | 148 | 151
Completed | 121 | 115
Not Completed | 30 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mycophenolate Mofetil + Sirolimus | Mycophenolate Mofetil + Cyclosporine or Tacrolimus | Total
Number analyzed (Participants) | 148 | 151 | 299
Age Continuous [Mean (Standard Deviation); unit: years] — Intent-to-treat population
  years | 48.7 (12.90) | 48.7 (12.70) | 48.7 (12.80)
Sex: Female, Male [Count of Participants; unit: Participants] — Intent-to-treat population
  Participants
    Female | 55 | 55 | 110
    Male | 93 | 96 | 189

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Glomerular Filtration Rate From Baseline to Month 12
Description: The primary efficacy endpoint was mean percent change in renal function from baseline to 12 months postrandomization, as measured by Glomerular Filtration Rate utilizing renal clearance of cold iothalamate.
  percent change= [(Glomerular Filtration Rate at Month 12-Glomerular Filtration Rate at baseline)/Glomerular Filtration Rate at baseline]*100 percent.
Time Frame: baseline to 12 months
Population: Intent-to-treat population. Analysis population (AP) at Baseline: Mycophenolate mofetil (MMF) + sirolimus = 148, MMF + cyclosporine or tacrolimus (CNI) = 151; AP at Month 12: MMF+sirolimus = 120, MMF+CNI = 111.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Mycophenolate Mofetil + Sirolimus | Mycophenolate Mofetil + Cyclosporine or Tacrolimus
Number analyzed (Participants) | 148 | 151
percent change
  Baseline | 59.5 (23.86) | 58.8 (26.06)
  Mean Percent Change from Baseline at Month 12 | 24.4 (70.00) | 5.2 (56.33)
Statistical Analysis 1: Comparison: Mycophenolate Mofetil + Sirolimus vs Mycophenolate Mofetil + Cyclosporine or Tacrolimus; The primary analysis tested the null hypothesis that mean percent change from baseline to 12 months for Group 1 (mycophenolate mofetil + sirolimus) was equal to that for Group 2 (mycophenolate mofetil + cyclosporine or tacrolimus) based on the intent-to-treat population; Test type: Superiority or Other; p = 0.012, ANCOVA — P value comparing the treatment groups calculated using ANCOVA model treatment and baseline calcineurin inhibitor (cyclosporine or tacrolimus) as factors and baseline measurement and time from transplant to randomization as covariates; Median Difference (Net) = 18.7, 95% CI [4.2 to 33.2]

2. Secondary Outcome: Mean Percent Change in Glomerular Filtration Rate From Baseline to Month 24
Description: A secondary efficacy endpoint was mean percent change in renal function from baseline to 24 months postrandomization, as measured by Glomerular Filtration Rate utilizing renal clearance of cold iothalamate.
  percent change= [(Glomerular Filtration Rate at Month 24-Glomerular Filtration Rate at baseline)/Glomerular Filtration Rate at baseline]*100 percent.
Time Frame: Baseline to 24 months
Population: Intent-to-treat population. Analysis population (AP) at Baseline: Mycophenolate mofetil (MMF) + sirolimus = 148, MMF + cyclosporine or tacrolimus (CNI) = 151; AP at Month 24: MMF+sirolimus = 115, MMF+CNI = 105.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Mycophenolate Mofetil + Sirolimus | Mycophenolate Mofetil + Cyclosporine or Tacrolimus
Number analyzed (Participants) | 148 | 151
percent change
  Baseline | 59.5 (23.86) | 58.8 (26.06)
  Percent Change from Baseline at Month 24 | 8.6 (55.32) | 3.4 (67.28)
Statistical Analysis 1: Comparison: Mycophenolate Mofetil + Sirolimus vs Mycophenolate Mofetil + Cyclosporine or Tacrolimus; Test type: Superiority or Other; p = 0.543, ANCOVA — P value comparing the treatment groups calculated using ANCOVA model treatment and baseline calcineurin inhibitor (cyclosporine or tacrolimus) type as factors and baseline measurement and time from transplant to randomization as covariates; Mean Difference (Net) = 4.3, 95% CI [-9.6 to 18.2]

3. Secondary Outcome: Mean Percent Change in Serum Creatinine From Baseline to Months 6, 12, and 24
Description: Renal allograft function determined by mean percent change from baseline in serum creatinine by treatment group at 6, 12, and 24 months postrandomization.
  percent change= [(serum creatinine at Month t-serum creatinine at baseline)/serum creatinine at baseline]*100 percent, where t=6, 12, and 24 months postrandomization.
Time Frame: baseline, 6, 12, and 24 months
Population: Intent-to-treat population. Analysis population (AP) at Baseline: Mycophenolate mofetil (MMF) + sirolimus = 148, MMF + cyclosporine or tacrolimus (CNI) = 151; AP at Month 6: MMF+sirolimus = 117, MMF+CNI = 130; AP at Month 12: MMF+sirolimus = 124, MMF+CNI = 123; AP at Month 24: MMF+sirolimus = 120, MMF+CNI = 116.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Mycophenolate Mofetil + Sirolimus | Mycophenolate Mofetil + Cyclosporine or Tacrolimus
Number analyzed (Participants) | 148 | 151
percent change
  Baseline | 121.1 (29.96) | 124.4 (37.87)
  Percent Change from Baseline at Month 6 | -3.7 (18.78) | 6.6 (34.61)
  Percent Change from Baseline at Month 12 | 6.0 (57.81) | 20.4 (92.81)
  Percent Change from Baseline at Month 24 | 6.1 (59.84) | 30.8 (114.23)
Statistical Analysis 1: Comparison: Mycophenolate Mofetil + Sirolimus vs Mycophenolate Mofetil + Cyclosporine or Tacrolimus; 6 months; Test type: Superiority or Other; p = 0.003, ANCOVA — P value comparing the two treatment groups is calculated using ANCOVA with treatment and baseline calcineurin inhibitor type (cyclosporine or tacrolimus) as factors, and baseline measurement and time from transplant to randomization as covariates; Median Difference (Net) = -10.8, 95% CI [-17.9 to -3.7]
Statistical Analysis 2: Comparison: Mycophenolate Mofetil + Sirolimus vs Mycophenolate Mofetil + Cyclosporine or Tacrolimus; 12 months; Test type: Superiority or Other; p = 0.108, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -16.0, 95% CI [-35.4 to 3.5]
Statistical Analysis 3: Comparison: Mycophenolate Mofetil + Sirolimus vs Mycophenolate Mofetil + Cyclosporine or Tacrolimus; 24 months; Test type: Superiority or Other; p = 0.039, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -24.4, 95% CI [-47.7 to -1.2]

4. Secondary Outcome: Mean Percent Change in Calculated Creatinine Clearance From Baseline to Months 6, 12, and 24
Description: Renal allograft function determined by mean percent change from baseline in calculated creatinine clearance (Cockroft and Gault method) by treatment group at 6, 12, and 24 months postrandomization.
  percent change= [(calculated creatinine clearance at Month t - calculated creatinine clearance at baseline)/calculated creatinine clearance at baseline]*100 percent, where t=6, 12, and 24 months postrandomization
Time Frame: baseline 6, 12, and 24 months
Population: Intent-to-treat population. Analysis population (AP) at Baseline: Mycophenolate mofetil (MMF) + sirolimus = 148, MMF + cyclosporine or tacrolimus (CNI) = 151; AP at Month 6: MMF+sirolimus = 117, MMF+CNI = 129; AP at Month 12: MMF+sirolimus = 124, MMF+CNI = 123; AP at Month 24: MMF+sirolimus = 120, MMF+CNI = 116.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Mycophenolate Mofetil + Sirolimus | Mycophenolate Mofetil + Cyclosporine or Tacrolimus
Number analyzed (Participants) | 148 | 151
percent change
  Baseline | 59.7 (16.85) | 60.5 (19.97)
  Percent Change from Baseline at Month 6 | 7.0 (19.54) | -1.7 (17.22)
  Percent Change from Baseline at Month 12 | 4.4 (24.38) | -2.3 (25.09)
  Percent Change from Baseline at Month 24 | 4.7 (27.58) | -4.2 (27.66)
Statistical Analysis 1: Comparison: Mycophenolate Mofetil + Sirolimus vs Mycophenolate Mofetil + Cyclosporine or Tacrolimus; 6 months; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 8.7, 95% CI [4.1 to 13.3]
Statistical Analysis 2: Comparison: Mycophenolate Mofetil + Sirolimus vs Mycophenolate Mofetil + Cyclosporine or Tacrolimus; 12 months; Test type: Superiority or Other; p = 0.029, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 6.9, 95% CI [0.7 to 13.1]
Statistical Analysis 3: Comparison: Mycophenolate Mofetil + Sirolimus vs Mycophenolate Mofetil + Cyclosporine or Tacrolimus; 24 months; Test type: Superiority or Other; p = 0.015, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 8.8, 95% CI [1.7 to 15.9]

5. Secondary Outcome: Mean Percent Change in Calculated Glomerular Filtration Rate From Baseline to Months 6, 12, and 24 (Nankivell Equation)
Description: Renal allograft function determined by mean percent change from baseline in calculated Glomerular Filtration Rate (Nankivell equation) by treatment group at 6, 12, and 24 months postrandomization.
  percent change= [(calculated Glomerular Filtration Rate at Month t - calculated Glomerular Filtration Rate at baseline)/calculated Glomerular Filtration Rate at baseline]*100 percent, where t=6, 12, and 24 months postrandomization.
Time Frame: baseline, 6, 12, and 24 months
Population: Intent-to-treat population. Analysis population (AP) at Baseline: Mycophenolate mofetil (MMF) + sirolimus = 148, MMF + cyclosporine or tacrolimus (CNI) = 151; AP at Month 6: MMF+sirolimus = 117, MMF+CNI = 130; AP at Month 12: MMF+sirolimus = 123, MMF+CNI = 123; AP at Month 24: MMF+sirolimus = 120, MMF+CNI = 116.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Mycophenolate Mofetil + Sirolimus | Mycophenolate Mofetil + Cyclosporine or Tacrolimus
Number analyzed (Participants) | 148 | 151
percent change
  Baseline | 71.3 (13.82) | 72.7 (16.2)
  Percent Change from Baseline at Month 6 | 8.3 (19.57) | -0.5 (15.98)
  Percent Change from Baseline at Month 12 | 5.2 (25.33) | -0.9 (23.42)
  Percent Change from Baseline at Month 24 | 6.5 (28.43) | -1.8 (27.31)
Statistical Analysis 1: Comparison: Mycophenolate Mofetil + Sirolimus vs Mycophenolate Mofetil + Cyclosporine or Tacrolimus; 6 months; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 8.5, 95% CI [4.2 to 12.9]
Statistical Analysis 2: Comparison: Mycophenolate Mofetil + Sirolimus vs Mycophenolate Mofetil + Cyclosporine or Tacrolimus; 12 months; Test type: Superiority or Other; p = 0.059, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 5.8, 95% CI [-0.2 to 11.9]
Statistical Analysis 3: Comparison: Mycophenolate Mofetil + Sirolimus vs Mycophenolate Mofetil + Cyclosporine or Tacrolimus; 24 months; Test type: Superiority or Other; p = 0.036, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 7.5, 95% CI [0.5 to 14.5]

ADVERSE EVENTS:
Description: Safety population. Three patients (38957/143, 38960/077, 38960/082) who were randomized to the Mycophenolate mofetil + sirolimus group did not switch to sirolimus after randomization and were included in the Mycophenolate Mofetil + cyclosporine or tacrolimus group for safety. These patients were excluded from the ITT population.
Arm/Group | Mycophenolate Mofetil + Sirolimus | Mycophenolate Mofetil + Cyclosporine or Tacrolimus
Serious Adverse Events (participants affected / at risk) | 60/148 | 64/153
Other Adverse Events (participants affected / at risk) | 147/148 | 148/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mycophenolate Mofetil + Sirolimus (N=148) | Mycophenolate Mofetil + Cyclosporine or Tacrolimus (N=153)
Pneumonia (Infections and infestations) | 14 | 9
Urinary Tract Infection (Infections and infestations) | 5 | 8
Pyelonephritis (Infections and infestations) | 4 | 3
Cellulitis (Infections and infestations) | 4 | 1
Urosepsis (Infections and infestations) | 3 | 2
Gastroenteritis (Infections and infestations) | 1 | 1
Gangrene (Infections and infestations) | 2 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 2
Osteomyelitis (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 2
Viral Infection (Infections and infestations) | 1 | 1
Appendicitis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 2
Bacterial Diarrhoea (Infections and infestations) | 1 | 0
BK Virus Infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Catheter Related Infection (Infections and infestations) | 0 | 1
Coccidioidomycosis (Infections and infestations) | 0 | 1
Diarrhoea Infectious (Infections and infestations) | 1 | 0
Ear Infection (Infections and infestations) | 1 | 0
Epstein-Barr Virus Infection (Infections and infestations) | 1 | 0
Escherichia Bacteraemia (Infections and infestations) | 0 | 1
Gastroenteritis Clostridial (Infections and infestations) | 1 | 0
Infected Skin Ulcer (Infections and infestations) | 1 | 0
Liver Abscess (Infections and infestations) | 1 | 0
Lung Abscess (Infections and infestations) | 1 | 0
Nocardiosis (Infections and infestations) | 1 | 0
Perinephric Abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal Abscess (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 1 | 0
Chest Pain (General disorders) | 4 | 3
Pyrexia (General disorders) | 4 | 3
Asthenia (General disorders) | 0 | 1
Chest Discomfort (General disorders) | 0 | 1
Hyperthermia (General disorders) | 0 | 1
Impaired Healing (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Gastritis (Gastrointestinal disorders) | 2 | 0
Diabetic Gastroparesis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus Paralytic (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1
Mouth Haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Retroperitoneal Haematoma (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 2
Focal Segmental Glomerulosclerosis (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 1 | 0
Urinary Tract Disorder (Renal and urinary disorders) | 2 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 3 | 1
Hypertensive Emergency (Vascular disorders) | 1 | 1
Peripheral Ischaemia (Vascular disorders) | 1 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Venous Stenosis (Vascular disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 1
Angina Unstable (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Supraventricular Tachyarrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Blood Creatinine Increased (Investigations) | 2 | 3
Blood Glucose Increased (Investigations) | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Haematuria (Injury, poisoning and procedural complications) | 0 | 1
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hungry Bone Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neuropathic Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 2
Brain Stem Infarction (Nervous system disorders) | 0 | 1
Cervical Cord Compression (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Intracranial Aneurysm (Nervous system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Haemolytic Uraemic Syndrome (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Knee Arthroplasty (Surgical and medical procedures) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Neuropathic Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 1
Serum Sickness (Immune system disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Breast Oedema (Reproductive system and breast disorders) | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 1
Normal Newborn (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Staphylococcal Bacteraemia (Infections and infestations) | 1 | 0
Cryptosporidiosis Infection (Infections and infestations) | 1 | 0
Groin Abscess (Infections and infestations) | 0 | 1
Benign Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute Prerenal Failure (Renal and urinary disorders) | 1 | 0
Urethral Stenosis (Renal and urinary disorders) | 1 | 0
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Open Reduction of Fracture (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mycophenolate Mofetil + Sirolimus (N=148) | Mycophenolate Mofetil + Cyclosporine or Tacrolimus (N=153)
Urinary Tract Infection (Infections and infestations) | 22 | 33
Upper Respiratory Tract Infection (Infections and infestations) | 21 | 19
Nasopharyngitis (Infections and infestations) | 13 | 16
Pneumonia (Infections and infestations) | 14 | 12
BK Virus Infection (Infections and infestations) | 0 | 9
Diarrhoea (Gastrointestinal disorders) | 51 | 50
Nausea (Gastrointestinal disorders) | 17 | 10
Vomiting (Gastrointestinal disorders) | 14 | 12
Abdominal Pain (Gastrointestinal disorders) | 9 | 14
Mouth Ulceration (Gastrointestinal disorders) | 21 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 8
Hyperlipidaemia (Metabolism and nutrition disorders) | 44 | 20
Hypokalaemia (Metabolism and nutrition disorders) | 20 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 9
Hypercholesterolaemia (Metabolism and nutrition disorders) | 9 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 9
Hypoglycaemia (Metabolism and nutrition disorders) | 8 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 8
Oedema Peripheral (General disorders) | 42 | 20
Fatigue (General disorders) | 15 | 12
Pyrexia (General disorders) | 15 | 12
Oedema (General disorders) | 10 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 11
Back Pain (Musculoskeletal and connective tissue disorders) | 15 | 6
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 12 | 9
Osteopenia (Musculoskeletal and connective tissue disorders) | 8 | 7
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 | 8
Osteoporosis (Musculoskeletal and connective tissue disorders) | 9 | 2
Blood Creatinine Increased (Investigations) | 14 | 31
Weight Increased (Investigations) | 7 | 8
Leukopenia (Blood and lymphatic system disorders) | 36 | 29
Anaemia (Blood and lymphatic system disorders) | 25 | 17
Polycythaemia (Blood and lymphatic system disorders) | 2 | 9
Neutropenia (Blood and lymphatic system disorders) | 2 | 7
Acne (Skin and subcutaneous tissue disorders) | 12 | 7
Rash (Skin and subcutaneous tissue disorders) | 8 | 7
Skin Ulcer (Skin and subcutaneous tissue disorders) | 8 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 16
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 0
Headache (Nervous system disorders) | 11 | 10
Dizziness (Nervous system disorders) | 8 | 8
Tremor (Nervous system disorders) | 1 | 14
Hypertension (Vascular disorders) | 30 | 25
Proteinuria (Renal and urinary disorders) | 18 | 6
Haematuria (Renal and urinary disorders) | 7 | 2
Insomnia (Psychiatric disorders) | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.